CLINICAL TRIAL: NCT04090424
Title: A Pivotal Study to Assess the Safety and Effectiveness of NovoSorb® Biodegradable Temporizing Matrix (BTM) in the Treatment of Severe Burn Skin Injuries
Brief Title: Assessment of Safety and Effectiveness of NovoSorb® BTM in Severe Burns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PolyNovo Biomaterials Pty Ltd. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-003
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NovoSorb BTM (Experimental): Application of NovoSorb BTM to study lesions
  Interventions: Device: NovoSorb BTM
- Standard of Care (Active Comparator): Application of the institution's standard of care to study lesions.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: NovoSorb BTM — NovoSorb BTM comprises a completely synthetic, sterile, integrating dermal component (porous biodegradable polyurethane foam) and a temporary epidermal barrier component (a nonbiodegradable polyurethane sealing membrane). These layers are adhered with a biodegradable polyurethane bonding layer. BTM will be implanted and fixed into position to close a debrided burn wound. After a period of integration, the sealing membrane is removed and a split skin graft is applied.
  Arms: NovoSorb BTM
Procedure: Standard of Care — Burn wounds will be treated using the institution's standard of care, e.g. primary skin grafting, cadaveric allograft followed by skin grafting.
  Arms: Standard of Care

SUMMARY:
This is a multi-center, pivotal study to assess the safety and effectiveness of a new method of treating severe burns using NovoSorb® Biodegradable Temporizing Matrix (BTM).

DETAILED DESCRIPTION:
This is a multi-center, pivotal study to assess the safety and effectiveness of a new method of treating severe burns using NovoSorb® Biodegradable Temporizing Matrix (BTM). A comparison will be made between burn wounds treated with BTM and the institution's standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent directly or via legal representative prior to any clinical study procedures being performed
2. Willing to comply with all study procedures and expects to be available for the duration of the study
3. Male and females ≥ 18 years of age and ≤ 75 years of age
4. Patients with deep dermal or full thickness burns between 3% and 60%, inclusive, of their total body surface area (TBSA).

   Types of burns include the following:
   * Scalding including from hot water, cooking oil, grease
   * Flame
   * Flash
   * Contact
5. Subjects who have staged surgical procedures planned e.g., one procedure to excise the burn injury and a later procedure to prepare the wound bed and apply an autologous skin graft.
6. The minimum total area across all lesions to have NovoSorb® BTM applied is 3% TBSA
7. Females, who are non-pregnant, naturally postmenopausal, or who agree to use effective contraceptive methods throughout the course of the study.

Exclusion Criteria:

1. Has a known hypersensitivity to polyurethane
2. Only a non-burn injury has been experienced by the subject including soft-tissue degloving and friction burn/crush, i.e., road rash
3. Multiple traumas, i.e., significant traumatic injury to a solid organ in addition to skin
4. Presence of a medical condition with a life expectancy of less than 12 months, such as advanced malignancy
5. Presence of a medical condition that might interfere with treatment evaluation; or require a change in therapy including but not limited to, significant immune deficiency, or skin or vascular diseases in the area of the wound
6. For females - has known or suspected pregnancy, planned pregnancy, or during lactation
7. Has exposure to any other investigational agent within the last 6 months
8. Has exposure to any other treatment/device that will interfere with NovoSorb® BTM integration
9. Anticipated inability to perform wound care and follow-up procedures
10. Anticipates of a level of non-compliance
11. The use of off-label treatments for full-thickness / deep-dermal burns is not permitted
12. Clinical signs of wound infection at areas to be potentially treated using NovoSorb® BTM that in the opinion of the investigator may compromise safety and study objectives
13. The use of NovoSorb® BTM on the face and in the perineum area is not permitted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of study lesions in both groups with complete wound closure after skin grafting | 4 weeks after skin grafting
  Assessment of clinical outcome by wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Wagstaff, MBBS, PhD, Study Director — Royal Adelaide Hospital, Adelaide SA 5000. Australia
Locations (26):
- United States (23):
  - Valleywise Health, Phoenix, Arizona
  - Southern California Regional Burn Center at LAC+USC, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - Loyola University of Chicago, Maywood, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University Medical Center, New Orleans, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York Presbyterian Weill Cornell Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Akron Children's Hospital, Burn Center, Akron, Ohio
  - The Ohio State University/ Wexner Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - UW Health University Hospital, Madison, Wisconsin
- India (3):
  - Bembde Hospital, Aurangabad, Maharashtra
  - National Burns Centre, Mumbai, Maharashtra
  - Ganga Medical Centre and Hospitals PVT Ltd, Coimbatore, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.polynovo.com.au/